CLINICAL TRIAL: NCT05141123
Title: A Physician-initiated, International, Multi-center, Retrospective and Prospective, Observational Registry of Patients Treated by Preloaded Fenestrated Stent-graft Designs for Complex Endovascular Aortic Procedures
Brief Title: Registry of Patients Treated by Preloaded Fenestrated Stent-graft Designs for Complex Endovascular Aortic Procedures
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Prof, IRCCS San Raffaele
Other Study IDs: Preloaded Registry
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Renal Aneurysm; Aneurysm Thoracic; Aneurysm Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preloaded Fenestrated Stent-graft Designs for Endovascular Aortic Procedures: Patients presenting with an acute (up to two weeks from the onset) and subacute (between 3 and 12 weeks from the onset) type B dissection with a proximal suitable non-dissected landing zone in the aortic arch or descending thoracic aorta (supra-aortic trunks debranching may be employed to obtain an adequate proximal landing zone)
  Interventions: Procedure: Complex Endovascular Aortic Procedures treated by Preloaded Fenestrated Stent-graft Designs for

INTERVENTIONS:
Procedure: Complex Endovascular Aortic Procedures treated by Preloaded Fenestrated Stent-graft Designs for — Evaluate the outcomes of the preloaded stent-graft design (PLD) in the routine treatment of para-renal and thoraco-abdominal aneurysms

SUMMARY:
The aim of the study is to evaluate the outcomes of the preloaded stent-graft design (PLD) in the routine treatment of para-renal and thoraco-abdominal aneurysms. Results and postoperative events are reported in accordance with the current reporting standards for endovascular aortic repair prepared and revised by the Ad Hoc Committee for Standardized Reporting Practices in Vascular Surgery of The Society for Vascular Surgery/American Association for Vascular Surgery.

The Registry will include approximately 300 patients treated from January 2015 to May 2021 (retrospective arm) and June 2021 to June 2023 (perspective arm) for the routine treatment of para-renal and thoraco-abdominal aneurysms. To reach 300 patients, the enrollments can be extended until June 2026.

ELIGIBILITY:
Inclusion Criteria:

-Patients presenting with an acute (up to two weeks from the onset) and subacute (between 3 and 12 weeks from the onset) type B dissection with a proximal suitable non-dissected landing zone in the aortic arch or descending thoracic aorta (supra-aortic trunks debranching may be employed to obtain an adequate proximal landing zone

Exclusion Criteria:

* Anatomy requiring sealing in the distal descending thoracic aorta may not be appropriate for a 50 cm sheath due to the risk of it being too short and the graft not reaching the intended landing zone;
* Celiac trunk or superior mesenteric branch design that makes the graft excessively long;
* Inability or refusal to give informed consent;
* Simultaneously participating in another investigative device or drug study;
* Frank rupture;
* Systemic infection (eg, sepsis);
* Allergy to stainless steel, polyester, solder (tin, silver), polypropylene, nitinol, or gold;
* Untreatable reaction to contrast, which, in the opinion of the investigator, cannot be adequately premedicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include approximately 300 patients treated from January 2015 to May 2021 (retrospective arm) and June 2021 to June 2023 (perspective arm) for the routine treatment of para-renal and thoraco-abdominal aneurysms. To reach 300 patients, the enrollments can be extended until June 2026.
Sampling Method: Non-Probability Sample
Enrollment: 741 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Clinical success | 30 days
  absence of death, type I/III endoleak, graft infection/thrombosis, aneurysm expansion and/or rupture, conversion to open repair, or new treatment-related thoraco-abdominal pathologies

CONTACTS AND LOCATIONS:
Locations (19):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Memorial Center for Complex Aortic Disease, Worcester, Massachusetts
  - Southwestern Medical Center, Dallas, Dallas, Texas
  - McGovern Medical School, Houston, Texas
  - University of Washington Seatle, Seattle, Washington
- Copenhagen Aortic Center, Copenhagen, Denmark
- France (4):
  - Centre Hospitalier Universitaire, Lille
  - Timone Hospital Marseille, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Aortic Centre Marie Lannelongue, Groupe Hospitalier Paris Saint Joseph, Université Paris Saclay, Paris
- Germany (3):
  - Hamburg Aortic Center, Hamburg
  - Ludwig Maximilian University Hospital, Munich
  - St. Franziskus Hospital, Münster
- Policlinico S. Orsola Malpighi, Bologna, Italy
- Hospital Doctor Peset, Valencia, Spain
- Sweden (2):
  - Vascular Center Malmö, Skåne University Hospital, Malmo
  - Department of Surgical Sciences, Vascular Surgery, Uppsala University, Uppsala
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Kings College, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberg RK, West K, Pfaff K, Foster J, Skender D, Haulon S, Sereika J, Geiger L, Lyden SP, Clair D, Svensson L, Lytle B. Beyond the aortic bifurcation: branched endovascular grafts for thoracoabdominal and aortoiliac aneurysms. J Vasc Surg. 2006 May;43(5):879-86; discussion 886-7. doi: 10.1016/j.jvs.2005.11.063. PMID 16678676
- [Background] Mohabbat W, Greenberg RK, Mastracci TM, Cury M, Morales JP, Hernandez AV. Revised duplex criteria and outcomes for renal stents and stent grafts following endovascular repair of juxtarenal and thoracoabdominal aneurysms. J Vasc Surg. 2009 Apr;49(4):827-37; discussion 837. doi: 10.1016/j.jvs.2008.11.024. Epub 2009 Feb 23. PMID 19233600
- [Background] Manning BJ, Harris PL, Hartley DE, Ivancev K. Preloaded fenestrated stent-grafts for the treatment of juxtarenal aortic aneurysms. J Endovasc Ther. 2010 Aug;17(4):449-55. doi: 10.1583/10-3024.1. PMID 20681756
- [Background] Kitagawa A, Greenberg RK, Eagleton MJ, Mastracci TM. Zenith p-branch standard fenestrated endovascular graft for juxtarenal abdominal aortic aneurysms. J Vasc Surg. 2013 Aug;58(2):291-300. doi: 10.1016/j.jvs.2012.12.087. Epub 2013 Apr 20. PMID 23611709
- [Background] Bisdas T, Donas KP, Torsello G, Austermann M. Technical assessment of the preloaded fenestrated stent-graft in the management of pararenal aortic aneurysms. J Endovasc Ther. 2013 Aug;20(4):461-8. doi: 10.1583/13-4310.1. PMID 23914852